CLINICAL TRIAL: NCT01346592
Title: A Phase III, Observer-Blind, Randomized, Multi-center Study to Evaluate the Safety, Tolerability, and Immunogenicity of Fluad and Agriflu Compared to the Non-adjuvanted Trivalent Influenza Vaccine Fluzone in Children 6 to < 72 Months of Age
Brief Title: Safety, Tolerability, and Immunogenicity of the Adjuvanted Trivalent Subunit Influenza Vaccine and the Non-Adjuvanted Trivalent Subunit Influenza Vaccine Compared to the Non-Adjuvanted Trivalent Split Influenza Vaccine in Children 6 to < 72 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V70_29
Record Dates: First submitted 2011-04-30; First posted 2011-05-03 (Estimated); Results first posted 2014-05-06 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Influenza Disease
Keywords: Adjuvanted Trivalent Subunit Influenza Vaccine; vaccine; influenza; adjuvant; MF-59; pediatric
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; fluad vaccine

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- aTIV (6 to <72 months) (Active Comparator): Subjects received an investigational MF59-adjuvanted trivalent influenza vaccine (aTIV), subjects aged between 6 to <36 months received two doses of 0.25 mL each, while subjects aged ≥36 months received two doses of 0.5 mL each, at Days 1 & 29
  Interventions: Biological: MF59-adjuvanted trivalent influenza vaccine (aTIV)
- Comparator TIV (6 to <72 months) (Active Comparator): Subjects received a licensed comparator trivalent split influenza vaccine (comparator TIV), subjects aged between 6 to <36 months received two doses of 0.25 mL each, while subjects aged ≥36 months received two doses of 0.5 mL each, at Days 1 & 29
  Interventions: Biological: Licensed comparator trivalent split influenza vaccine (comparator TIV)
- TIV (6 to <72 months) (Active Comparator): Subjects received an investigational trivalent split influenza vaccine (TIV), subjects aged between 6 to <36 months received two doses of 0.25 mL each, while subjects aged ≥36 months received two doses of 0.5 mL each, at Days 1 & 29
  Interventions: Biological: Trivalent split influenza vaccine (TIV)

INTERVENTIONS:
Biological: Trivalent split influenza vaccine (TIV)
  Other Names: Agriflu
  Arms: TIV (6 to <72 months)
Biological: MF59-adjuvanted trivalent influenza vaccine (aTIV)
  Other Names: Fluad
  Arms: aTIV (6 to <72 months)
Biological: Licensed comparator trivalent split influenza vaccine (comparator TIV)
  Other Names: Fluzone
  Arms: Comparator TIV (6 to <72 months)

SUMMARY:
This Study Aims to Evaluate the Safety, Tolerability, and Immunogenicity of the Adjuvanted Trivalent Subunit Influenza Vaccine and the Non-Adjuvanted Trivalent Subunit Influenza Vaccine Compared to the Non-Adjuvanted Trivalent Split Influenza Vaccine in Children 6 to < 72 Months of Age.

ELIGIBILITY:
Inclusion Criteria:

1.Children 6 months to 72 months of age.

Exclusion Criteria:Children

1. Who had been hospitalized at the time of enrollment
2. Who had any serious reaction or hypersensitivity to any vaccine component, eggs, or chicken protein
3. Who had known impairment of the immune function
4. Who had fever interfering with normal daily activities at the time of enrollment
5. Who had received licensed vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in the study
6. Concomitant participation in another clinical study
7. Who had surgery planned during the study period that in the investigator's opinion would have interfered with the study visits schedule.

Ages: 6 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6104 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (34):
- Argentina (8):
  - 401 Paideia Jeronimo Salguero 2835 Piso 1, Buenos Aires
  - 402 Hospital de Ninos Gallo 130, Buenos Aires
  - 403 Instituto Medico Rio Cuarto Hipolito Yrigoyen 1020, Córdoba
  - 405 Hospital Pediatrico Nino Jesus Castro Barros 650, Córdoba
  - 406 Hospital Nostra Senora de la Misericordia Belgrano 1500, Córdoba
  - 407 Centro Pediatrico Caballito Directorio 1658, Cuidad Automa de Beunos Aires
  - 408 Centro de Salud 31 Serpa y Republica del Libano, Mendoza
  - 409 Centro de Salud 16 Alpatacal y Chile, Villa Nueva
- Australia (5):
  - 206 Vaccine and Immunology Research Trials Unit University Department of Paediatrics 2nd floor Clarence Reiger Bldg Womens and Childrens Hospital, Adelaide
  - 201 Royal Children Hospital Department of Respiratory Medicine, Herston
  - 205 Vaccine and Immunisation Research Group Murdoch Childrens Research Institute School Of Population Health, Level 5 207 Bouverie Saint
  - 202 Sydney Children Hospital Department of Immunology and Infectious Diseases, Randwick
  - 204 National Centre for Immunisation Research and Surveillance Kids Research Institute The Childrens Hospital at Westmead, Westmead
- Chile (2):
  - 502 Hospital Clinico Pontificia Universidad Catolica de Chile Marcoleta 357, Santiago
  - 503 Clinica Tabancura Av Tabancura 1185, Santiago
- Philippines (14):
  - 111 DLSHI deCastro De La Salle Health Sciences Institute DBB B Dasmarinas, Cavite
  - 106 Research Institute for Tropical Medicine Alabang Muntinlupa, City of Muntinlupa
  - 108 RITM Research Institute for Tropical Medicine Department of Health Compound FILINVEST Corporate City Alabang, City of Muntinlupa
  - 109 De La Salle Health Sciences Institute, Dbbb Dasmarinas Cavite
  - 110 De La Salle Health Sciences Institute, Dbbb Dasmarinas Cavite
  - 103 Philippine General Hospital Taft Avenue, Manila
  - 107 Philippine General Hospital Taft Avenue, Manila
  - 112 PGH Lim Philippine General Hospital Taft Avenue, Manila
  - 114 Philippine General Hospital Taft Avenue, Manila
  - 105 Mary Chiles General Hospital 667 Gastambide St Sampaloc Manila, Manila
  - 102 University of the East Ramon Magsaysay Memorial 64 Aurora Boulevard Barangay Dona Imelda, Quezon
  - 101 Philippine Childrens Medical Center Quezon Avenue cor Agham Road Quezon City, Quezon City
  - 104 Philippine Childrens Medical Center Quezon Avenue cor Agham Road Quezon City, Quezon City
  - 113 Philippine Childrens Medical Center Quezon Avenue cor Agham Road Quezon City, Quezon City
- South Africa (5):
  - 305 Worthwhile Clinical Trials Lakeview Hospital 1 Mowbray Avenue, Benoni
  - 304 Newgate Centre Suite 3, Johannesburg
  - 303 Emmed Research, Pretoria
  - 301 Perinatal HIV Research Unit, Baragwanath Hospital, Soweto
  - 302 Soweto Clinical Research, Soweto

REFERENCES:
- [Derived] Nolan T, Bravo L, Ceballos A, Mitha E, Gray G, Quiambao B, Patel SS, Bizjajeva S, Bock H, Nazaire-Bermal N, Forleo-Neto E, Cioppa GD, Narasimhan V. Enhanced and persistent antibody response against homologous and heterologous strains elicited by a MF59-adjuvanted influenza vaccine in infants and young children. Vaccine. 2014 Oct 21;32(46):6146-56. doi: 10.1016/j.vaccine.2014.08.068. Epub 2014 Sep 16. PMID 25223266

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 8 sites in Argentina, 5 sites in Australia, 2 sites in Chile, 12 sites in Philippines, and 5 sites in South Africa.
Pre-assignment Details: 4 of the enrolled subjects were not randomized hence were not included in the trial.
Period: Overall Study
Arm/Group | aTIV (6 to <72 Months) | Comparator TIV (6 to <72 Months) | TIV (6 to <72 Months)
Started | 3136 | 1478 | 1486
Completed | 2983 | 1389 | 1408
Not Completed | 153 | 89 | 78
Not completed — Lost to Follow-up | 62 | 29 | 29
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Death | 1 | 3 | 4
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 77 | 51 | 38
Not completed — Inappropriate enrollment | 3 | 1 | 1
Not completed — Administrative reason | 1 | 0 | 0
Not completed — Unable to Classify | 7 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | aTIV (6 to <72 Months) | Comparator TIV (6 to <72 Months) | TIV (6 to <72 Months) | Total
Number analyzed (Participants) | 3136 | 1478 | 1486 | 6100
Age, Continuous [Mean (Standard Deviation); unit: Months] | 37.1 (18.6) | 30.0 (16.9) | 30.2 (16.9) | 33.7 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1545 | 745 | 731 | 3021
  Male | 1591 | 733 | 755 | 3079

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Antibody Responses of aTIV With TIV and Comparator TIV in Terms of Geometric Mean Titers (GMTs) Against Homologous Strains
Description: The non-inferiority of Hemagglutination Inhibition (HI) antibody responses of aTIV compared to TIV and comparator TIV assessed in terms of post vaccination GMTs at three weeks after last vaccination against the three homologous vaccine strains.
Time Frame: Day 1, Day 50
Population: Analysis was done on the Per Protocol Set (PPS) i.e all subjects in the enrolled population who correctly received the study vaccine, provided evaluable serum samples at relevant time-points and had no major protocol violations as defined prior to unblinding.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- aTIV (6 to <72 Months): Subjects received an investigational MF59-adjuvanted trivalent influenza vaccine (aTIV), subjects aged between 6 to <36 months received two doses (Day 1 & 29) while subjects aged ≥36 months received one dose (at Day 1) of the vaccine
- Comparator TIV (6 to <72 Months): Subjects received a licensed comparator trivalent split influenza vaccine (comparator TIV), subjects aged between 6 to <36 months received two doses (Day 1 & 29) while subjects aged ≥36 months received one dose (at Day 1) of the vaccine
- TIV (6 to <72 Months): Subjects received an investigational trivalent split influenza vaccine (TIV), subjects aged between 6 to <36 months received two doses (Day 1 & 29) while subjects aged ≥36 months received one dose (Day 1) of the vaccine
Arm/Group | aTIV (6 to <72 Months) | Comparator TIV (6 to <72 Months) | TIV (6 to <72 Months)
Number analyzed (Participants) | 682 | 757 | 765
Titers
  H1N1 - Day 1 (N=681,757,765) | 28 [24 to 33] | 24 [21 to 28] | 27 [23 to 31]
  H1N1 - Day 50 (N=681,757,765) | 1537 [1382 to 1709] | 629 [567 to 698] | 480 [433 to 532]
  H3N2 - Day 1 | 40 [35 to 47] | 42 [36 to 49] | 44 [38 to 51]
  H3N2 - Day 50 | 1908 [1785 to 2040] | 1012 [948 to 1080] | 803 [752 to 857]
  B strain Day 1 | 9.87 [9.08 to 11] | 10 [9.41 to 11] | 10 [9.33 to 11]
  B strain Day 50 | 492 [450 to 537] | 160 [147 to 175] | 157 [144 to 171]
Statistical Analysis 1: Comparison: aTIV (6 to <72 Months) vs Comparator TIV (6 to <72 Months); Test type: Non-Inferiority or Equivalence — Noninferiority was established if the lower limit of the confidence interval of the day 50 ratio of GMTs was >0.667; GMT ratio (H1N1 strain) = 2.44, 97.6% CI 2-sided [2.06 to 2.9]
Statistical Analysis 2: Comparison: aTIV (6 to <72 Months) vs Comparator TIV (6 to <72 Months); Test type: Non-Inferiority or Equivalence — Noninferiority was established if the lower limit of the confidence interval of the day 50 ratio of GMTs was >0.667; GMT ratio (H3N2 strain) = 1.89, 97.6% CI 2-sided [1.69 to 2.1]
Statistical Analysis 3: Comparison: aTIV (6 to <72 Months) vs Comparator TIV (6 to <72 Months); Test type: Non-Inferiority or Equivalence — Noninferiority was established if the lower limit of the confidence interval of the day 50 ratio of GMTs was >0.667; GMT ratio (B strain) = 3.07, 97.6% CI 2-sided [2.66 to 3.54]
Statistical Analysis 4: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); Test type: Non-Inferiority or Equivalence — Noninferiority was established if the lower limit of the confidence interval of the day 50 ratio of GMTs was >0.667; GMT ratio (H1N1 strain) = 3.2, 97.6% CI 2-sided [2.7 to 3.8]
Statistical Analysis 5: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); Test type: Non-Inferiority or Equivalence — Noninferiority was established if the lower limit of the confidence interval of the day 50 ratio of GMTs was >0.667; GMT ratio (H3N2 strain) = 2.38, 97.6% CI 2-sided [2.14 to 2.65]
Statistical Analysis 6: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); Test type: Non-Inferiority or Equivalence — Noninferiority was established if the lower limit of the confidence interval of the day 50 ratio of GMTs was >0.667; GMT ratio (B strain) = 3.14, 97.6% CI 2-sided [2.72 to 3.62]

2. Primary Outcome: Comparison of Antibody Responses of aTIV With TIV and Comparator TIV in Terms of Percentage of Subjects Achieving Seroconversion or ≥4-fold Increase in HI Titers Against Homologous Strains
Description: The non-inferiority of HI antibody responses of aTIV compared to TIV and comparator TIV assessed in terms of percentage of subjects achieving seroconversion or ≥4-fold increase in HI titers at three weeks after last vaccination against the three homologous vaccine strains.
  Seroconversion defined as prevaccination HI titer <10 and postvaccination HI titer ≥40 or at least a 4-fold increase in HI titers from prevaccination HI titer ≥10.
Time Frame: Day 50
Population: Analysis was done on the PPS.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (6 to <72 Months) | Comparator TIV (6 to <72 Months) | TIV (6 to <72 Months)
Number analyzed (Participants) | 682 | 757 | 765
Percentage of subjects
  H1N1 - (N=680,757,765) | 92.9 [90.8 to 94.8] | 84.5 [81.8 to 87.1] | 79.4 [76.3 to 82.2]
  H3N2 | 96.5 [94.8 to 97.7] | 92.3 [90.2 to 94.1] | 89.4 [87 to 91.5]
  B strain | 98 [96.6 to 98.9] | 86 [83.3 to 88.4] | 84.6 [81.8 to 87.1]
Statistical Analysis 1: Comparison: aTIV (6 to <72 Months) vs Comparator TIV (6 to <72 Months); Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the lower bound of the confidence interval for day 50 vaccine group difference was >-10%; Group difference (H1N1 strain) = 9.09, 97.6% CI 2-sided [5.48 to 12.69]
Statistical Analysis 2: Comparison: aTIV (6 to <72 Months) vs Comparator TIV (6 to <72 Months); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Group difference (H3N2 strain) = 4.07, 97.6% CI 2-sided [1.58 to 6.55]
Statistical Analysis 3: Comparison: aTIV (6 to <72 Months) vs Comparator TIV (6 to <72 Months); Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the lower bound of the confidence interval for day 50 vaccine group difference was > -10%; Group difference (B strain) = 11.82, 97.6% CI 2-sided [8.72 to 14.92]
Statistical Analysis 4: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; Group difference (H1N1 strain) = 14.21, 97.6% CI 2-sided [10.3 to 18.13]
Statistical Analysis 5: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; Group difference (H3N2 strain) = 7.31, 97.6% CI 2-sided [4.47 to 10.14]
Statistical Analysis 6: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; Group difference (B strain) = 11.1, 97.6% CI 2-sided [8.11 to 14.1]

3. Primary Outcome: Comparison of Antibody Responses of TIV Versus Comparator TIV in Terms of Geometric Mean Titers (GMTs) Against Homologous Strains (6 to <36 Months)
Description: The non-inferiority of HI antibody responses of TIV to that of comparator TIV, in subjects aged 6 to <36 Months, assessed in terms of post vaccination GMTs at three weeks after last vaccination against the three homologous vaccine strains.
Time Frame: Day 1, Day 50
Population: Analysis was done on the PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- TIV (6 to <36months): Subjects received two doses of 0.25 mL each, of investigational trivalent split influenza vaccine (TIV), at Days 1 & 29
- Comparator TIV (6 to <36months): Subjects received two doses of 0.25 mL each, of the licensed trivalent split influenza vaccine (comparator TIV), at Days 1 & 29
Arm/Group | TIV (6 to <36months) | Comparator TIV (6 to <36months)
Number analyzed (Participants) | 642 | 635
Titers
  H1N1 - Day 1 | 23 [20 to 27] | 20 [17 to 23]
  H1N1 - Day 50 | 370 [328 to 419] | 487 [431 to 551]
  H3N2 - Day 1 | 29 [24 to 33] | 28 [24 to 33]
  H3N2 - Day 50 | 698 [650 to 749] | 912 [849 to 980]
  B strain Day 1 | 9.42 [8.63 to 10] | 9.42 [8.62 to 10]
  B -strain Day 50 | 144 [130 to 159] | 152 [138 to 168]
Statistical Analysis 1: Comparison: TIV (6 to <36months) vs Comparator TIV (6 to <36months); Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the lower bound of the confidence interval for day 50 GMT group ratios was >0.667; Group ratio (H1N1 strain) = 0.76, 97.4% CI 2-sided [0.62 to 0.93]
Statistical Analysis 2: Comparison: TIV (6 to <36months) vs Comparator TIV (6 to <36months); Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the lower bound of the confidence interval for day 50 GMT group ratios was >0.667; GMT ratio (H3N2 strain) = 0.77, 97.4% CI 2-sided [0.68 to 0.86]
Statistical Analysis 3: Comparison: TIV (6 to <36months) vs Comparator TIV (6 to <36months); Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the lower bound of the confidence interval for day 50 GMT group ratios was >0.667; GMT ratio (B strain) = 0.94, 97.4% CI 2-sided [0.8 to 1.11]

4. Primary Outcome: Comparison of Antibody Responses of TIV Versus Comparator TIV in Terms of Percentage of Subjects Achieving Seroconversion or ≥4-fold Increase in HI Titer Against Homologous Strains in Subjects 6 to <36 Months of Age
Description: The non-inferiority of HI antibody responses of TIV to that of the licensed comparator TIV assessed in terms of percentage of subjects achieving seroconversion or ≥4-fold increase in HI titers at three weeks after last vaccination against the three homologous vaccine strains.
Time Frame: Day 50
Population: Subjects aged 6 through <36 months of age - Per Protocol Set (PPS).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TIV (6 to <36months) | Comparator TIV (6 to <36months)
Number analyzed (Participants) | 642 | 635
Percentage of subjects
  H1N1 | 78.8 [75.5 to 81.9] | 84.1 [81 to 86.9]
  H3N2 | 89.9 [87.3 to 92.1] | 92.6 [90.3 to 94.5]
  B strain | 82.7 [79.6 to 85.6] | 85.5 [82.5 to 88.2]
Statistical Analysis 1: Comparison: TIV (6 to <36months) vs Comparator TIV (6 to <36months); Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the lower bound of the confidence interval for day 50 vaccine group differences was > -10%; Group difference (H1N1 strain) = -5.3, 97.4% CI 2-sided [-10.13 to -0.47]
Statistical Analysis 2: Comparison: TIV (6 to <36months) vs Comparator TIV (6 to <36months); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Group difference (H3N2 strain) = -2.84, 97.4% CI 2-sided [-6.16 to 0.5]
Statistical Analysis 3: Comparison: TIV (6 to <36months) vs Comparator TIV (6 to <36months); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Group difference (B strain) = -2.49, 97.4% CI 2-sided [-7.01 to 2]

5. Secondary Outcome: Comparison of Antibody Responses of aTIV With TIV and Comparator TIV in Terms of GMTs Against Homologous Strains (6 to <24 Months)
Description: The superiority of HI antibody responses, in subjects 6 to <24 months of age, of aTIV compared to TIV and comparator TIV assessed in terms of post vaccination GMTs at three weeks after last vaccination against the three homologous vaccine strains.
Time Frame: Day 1, Day 50
Population: Analysis was done on the Full Analysis Set (FAS) i.e all enrolled subjects who received study vaccination and provided serum samples.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- aTIV (6 to <24 Months): Subjects received two doses of 0.25 mL each, of the investigational MF59-adjuvanted trivalent split influenza vaccine (aTIV), at Days 1 & 29
- Comparator TIV (6 to <24 Months): Subjects received two doses of 0.25 mL each, of the licensed comparator trivalent split influenza vaccine (comparator TIV), at Days 1 & 29
- TIV (6 to <24 Months): Subjects received two doses of 0.25 mL each, of the investigational trivalent split influenza vaccine (TIV), at Days 1 & 29
Arm/Group | aTIV (6 to <24 Months) | Comparator TIV (6 to <24 Months) | TIV (6 to <24 Months)
Number analyzed (Participants) | 266 | 389 | 387
Titers
  H1N1 - Day 1 | 12 [9.52 to 14] | 9.87 [8.36 to 12] | 12 [9.95 to 14]
  H1N1 - Day 50 | 1080 [899 to 1297] | 298 [256 to 347] | 205 [176 to 238]
  H3N2 - Day 1 | 15 [12 to 19] | 15 [12 to 18] | 17 [14 to 21]
  H3N2 - Day 50 | 1709 [1536 to 1903] | 758 [694 to 828] | 552 [505 to 603]
  B strain Day 1 | 7.75 [6.83 to 8.78] | 8.18 [7.37 to 9.07] | 7.92 [7.14 to 8.79]
  B strain Day 50 | 616 [534 to 711] | 133 [118 to 149] | 112 [100 to 127]
Statistical Analysis 1: Comparison: aTIV (6 to <24 Months) vs Comparator TIV (6 to <24 Months); Superiority was concluded if the lower limit of the confidence interval for the day 50 vaccine group GMT ratios for at least 2 homologous strains was >1.5; Test type: Superiority or Other; GMT ratio (H1N1 strain) = 3.63, 95% CI 2-sided [2.86 to 4.6]
Statistical Analysis 2: Comparison: aTIV (6 to <24 Months) vs Comparator TIV (6 to <24 Months); superiority was concluded if the lower limit of the confidence interval of the day 50 vaccine group GMT ratios for at least 2 homologous strains was >1.5; Test type: Superiority or Other; GMT ratio (H3N2 strain) = 2.25, 95% CI 2-sided [1.96 to 2.59]
Statistical Analysis 3: Comparison: aTIV (6 to <24 Months) vs Comparator TIV (6 to <24 Months); [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; GMT ratio (B strain) = 4.64, 95% CI 2-sided [3.86 to 5.59]
Statistical Analysis 4: Comparison: aTIV (6 to <24 Months) vs TIV (6 to <24 Months); [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; GMT ratio (H1N1 strain) = 5.28, 95% CI 2-sided [4.16 to 6.7]
Statistical Analysis 5: Comparison: aTIV (6 to <24 Months) vs TIV (6 to <24 Months); [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; GMT ratio (H3N2 strain) = 3.1, 95% CI 2-sided [2.69 to 3.56]
Statistical Analysis 6: Comparison: aTIV (6 to <24 Months) vs TIV (6 to <24 Months); [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; GMT ratio (B strain) = 4.64, 95% CI 2-sided [3.86 to 5.59]

6. Secondary Outcome: Comparison of Antibody Responses of aTIV With TIV and Comparator TIV in Terms Percentage of Subjects Achieving Seroconversion or ≥4-fold Increase in HI Titer Against Homologous Strains (6 to <24 Months)
Description: The superiority of HI antibody responses, in subjects 6 to <24 months of age, of aTIV compared to TIV and comparator TIV assessed in terms of number of subjects achieving seroconversion at three weeks after last vaccination against the three homologous vaccine strains.
Time Frame: Day 50
Population: Analysis was done on the FAS
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (6 to <24 Months) | Comparator TIV (6 to <24 Months) | TIV (6 to <24 Months)
Number analyzed (Participants) | 266 | 389 | 387
Percentage of subjects
  H1N1 | 95.5 [92.3 to 97.7] | 85.1 [81.2 to 88.5] | 77.8 [73.3 to 81.8]
  H3N2 | 98.1 [95.7 to 99.4] | 95.6 [93.1 to 97.4] | 92.5 [89.4 to 94.9]
  B strain | 98.1 [95.7 to 99.4] | 85.4 [81.4 to 88.7] | 79.3 [75 to 83.3]
Statistical Analysis 1: Comparison: aTIV (6 to <24 Months) vs Comparator TIV (6 to <24 Months); superiority was concluded if the lower limit of the confidence interval of day 50 vaccine group difference,for at least 2 homologous strains, was >10%; Test type: Superiority or Other; Group difference (H1N1 strain) = 10.4, 95% CI 2-sided [6.1 to 14.7]
Statistical Analysis 2: Comparison: aTIV (6 to <24 Months) vs Comparator TIV (6 to <24 Months); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Group difference (H3N2 strain) = 2.5, 95% CI 2-sided [-0.12 to 5.1]
Statistical Analysis 3: Comparison: aTIV (6 to <24 Months) vs Comparator TIV (6 to <24 Months); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Group difference (B strain) = 12.8, 95% CI 2-sided [8.9 to 16.7]
Statistical Analysis 4: Comparison: aTIV (6 to <24 Months) vs TIV (6 to <24 Months); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Group difference (H1N1 strain) = 17.7, 95% CI 2-sided [12.9 to 22.6]
Statistical Analysis 5: Comparison: aTIV (6 to <24 Months) vs TIV (6 to <24 Months); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Group difference (H3N2 strain) = 5.6, 95% CI 2-sided [2.5 to 8.7]
Statistical Analysis 6: Comparison: aTIV (6 to <24 Months) vs TIV (6 to <24 Months); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Group difference (B strain) = 18.8, 95% CI 2-sided [14.4 to 23.1]

7. Secondary Outcome: Comparison of Antibody Responses of aTIV With TIV and Comparator TIV in Terms of GMTs Against Homologous Strains (6 to <72 Months)-FAS
Description: The superiority of HI antibody responses, in subjects 6 to <72 months of age, of aTIV compared to TIV and comparator TIV assessed in terms of post vaccination GMTs at three weeks after last vaccination against the three homologous vaccine strains.
Time Frame: Day 1, Day 50
Population: Analysis was done on the FAS
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | aTIV (6 to <72 Months) | Comparator TIV (6 to <72 Months) | TIV (6 to <72 Months)
Number analyzed (Participants) | 747 | 839 | 849
Titers
  H1N1 - Day 1 (N=746,839,849) | 29 [25 to 33] | 24 [21 to 28] | 27 [23 to 31]
  H1N1 - Day 50 (N=746,839,849) | 1519 [1372 to 1683] | 637 [577 to 704] | 473 [428 to 522]
  H3N2 - Day 1 | 41 [36 to 48] | 42 [37 to 49] | 44 [38 to 50]
  H3N2 - Day 50 | 1909 [1791 to 2035] | 1016 [954 to 1081] | 796 [748 to 847]
  B strain - Day 1 | 9.97 [9.2 to 11] | 10 [9.49 to 11] | 10 [9.33 to 11]
  B strain-Day 50 | 480 [441 to 523] | 164 [151 to 178] | 156 [144 to 169]
Statistical Analysis 1: Comparison: aTIV (6 to <72 Months) vs Comparator TIV (6 to <72 Months); [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; GMT Ratio (H1N1 strain) = 2.38, 95% CI 2-sided [2.07 to 2.75]
Statistical Analysis 2: Comparison: aTIV (6 to <72 Months) vs Comparator TIV (6 to <72 Months); [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; GMT Ratio (H3N2 strain) = 1.88, 95% CI 2-sided [1.72 to 2.06]
Statistical Analysis 3: Comparison: aTIV (6 to <72 Months) vs Comparator TIV (6 to <72 Months); [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; GMT Ratio (B strain) = 2.93, 95% CI 2-sided [2.6 to 3.3]
Statistical Analysis 4: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; GMT Ratio (H1N1 strain) = 3.21, 95% CI 2-sided [2.79 to 3.71]
Statistical Analysis 5: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; GMT Ratio (H3N2 strain) = 2.4, 95% CI 2-sided [2.19 to 2.62]
Statistical Analysis 6: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; GMT Ratio (B strain) = 3.08, 95% CI 2-sided [2.73 to 3.47]

8. Secondary Outcome: Comparison of Antibody Responses of aTIV With TIV and Comparator TIV in Terms of Percentage of Subjects Achieving Seroconversion or ≥4 Fold Increase in HI Titers Against Homologous Strains (6 to <72 Months)-FAS
Description: The superiority of HI antibody responses, in subjects 6 to <24 months of age, of aTIV compared to TIV and comparator TIV assessed in terms of number of subjects achieving seroconversion ≥4 fold increase in HI titers at three weeks after last vaccination against the three homologous vaccine strains.
Time Frame: Day 50
Population: Analysis was done on the FAS
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (6 to <72 Months) | Comparator TIV (6 to <72 Months) | TIV (6 to <72 Months)
Number analyzed (Participants) | 747 | 839 | 849
Percentage of subjects
  H1N1 | 92.8 [90.7 to 94.5] | 83.7 [81 to 86.1] | 78.8 [75.9 to 81.5]
  H3N2 | 96.4 [94.8 to 97.6] | 92.3 [90.2 to 94] | 89.8 [87.5 to 91.7]
  B strain | 97.5 [96.1 to 98.5] | 86.4 [83.9 to 88.7] | 84.5 [81.8 to 86.8]
Statistical Analysis 1: Comparison: aTIV (6 to <72 Months) vs Comparator TIV (6 to <72 Months); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Group difference (H1N1 strain) = 9.3, 95% CI 2-sided [6.3 to 12.4]
Statistical Analysis 2: Comparison: aTIV (6 to <72 Months) vs Comparator TIV (6 to <72 Months); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Group difference (H3N2 strain) = 3.9, 95% CI 2-sided [1.8 to 5.9]
Statistical Analysis 3: Comparison: aTIV (6 to <72 Months) vs Comparator TIV (6 to <72 Months); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Group difference (B strain) = 10.7, 95% CI 2-sided [8.1 to 13.3]
Statistical Analysis 4: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Group difference (H1N1 strain) = 14.4, 95% CI 2-sided [11.1 to 17.7]
Statistical Analysis 5: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); superiority was concluded if the lower bound of 95% CI of day 50 vaccine group difference,for at least 2 homologous strains, was >10%; Test type: Superiority or Other; Group difference (H3N2 strain) = 6.8, 95% CI 2-sided [4.5 to 9.1]
Statistical Analysis 6: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Group difference (B strain) = 10.9, 95% CI 2-sided [8.3 to 13.4]

9. Secondary Outcome: The HI GMTs Against Homologous Strains, by Vaccine Group
Description: The HI antibody titers against the three homologous strains following vaccination with either aTIV, licensed comparator or TIV, at three weeks and at six months after vaccination are reported as GMTs.
Time Frame: Day 1, Day 29, Day 50, Day 209
Population: Analysis was done on FAS (Persistence) i.e. all subjects in the enrolled population who actually received a study vaccination, and provided evaluable serum samples at all relevant timepoints and also at day 209.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | aTIV (6 to <72 Months) | Comparator TIV (6 to <72 Months) | TIV (6 to <72 Months)
Number analyzed (Participants) | 715 | 822 | 820
Titers
  H1N1 - Day 1 (N=714,822,820) | 28 [24 to 32] | 24 [20 to 27] | 27 [23 to 31]
  H1N1 - Day 29 | 647 [562 to 745] | 159 [139 to 182] | 170 [148 to 194]
  H1N1 - Day 50 (N=714,822,820) | 1507 [1358 to 1673] | 635 [575 to 702] | 475 [429 to 525]
  H1N1 - Day 209 (N=715,822,819) | 276 [246 to 311] | 97 [87 to 109] | 107 [96 to 120]
  H3N2 - Day 1 | 42 [36 to 48] | 43 [37 to 49] | 43 [38 to 50]
  H3N2 - Day 29 | 1087 [1004 to 1176] | 558 [517 to 602] | 453 [420 to 490]
  H3N2 - Day 50 | 1920 [1799 to 2050] | 1013 [952 to 1079] | 810 [760 to 862]
  H3N2 - Day 209 | 462 [423 to 505] | 277 [254 to 301] | 242 [222 to 263]
  B - Day 1 | 10 [9.29 to 11] | 10 [9.57 to 11] | 10 [9.34 to 11]
  B - Day 29 | 119 [106 to 134] | 58 [52 to 65] | 61 [54 to 68]
  B - Day 50 | 488 [447 to 532] | 166 [153 to 180] | 159 [146 to 173]
  B- Day 209 | 125 [114 to 136] | 57 [53 to 62] | 61 [56 to 66]

10. Secondary Outcome: Geometric Mean Ratio (GMR) of Post- Versus Pre-vaccination HI Titers Against Homologous Strains
Description: The GMR of post-vaccination versus pre-vaccination HI titers against homologous strains, three weeks (day 29/day 1; day 50/day 1)and six months (day 209/day 1) after vaccination with either aTIV, licensed comparator or TIV.
Time Frame: Day 29, Day 50, Day 209
Population: Analysis was done on FAS (Persistence)
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | aTIV (6 to <72 Months) | Comparator TIV (6 to <72 Months) | TIV (6 to <72 Months)
Number analyzed (Participants) | 715 | 822 | 820
Ratios
  H1N1, Day 29:Day 1 (N=714,822,820) | 27 [23 to 31] | 6.81 [5.94 to 7.81] | 7.13 [6.22 to 8.18]
  H1N1, Day 50:Day 1 (N=713,822,820) | 58 [51 to 67] | 27 [24 to 31] | 19 [17 to 21]
  H1N1, Day 209:Day 1 (N=714,822,819) | 11 [9.79 to 13] | 4.15 [3.68 to 4.69] | 4.37 [3.87 to 4.94]
  H3N2, Day 29:Day 1 | 29 [26 to 32] | 15 [14 to 16] | 12 [11 to 13]
  H3N2, Day 50:Day 1 (N=715,822,820) | 48 [43 to 54] | 25 [23 to 28] | 20 [18 to 22]
  H3N2, Day 209:Day 1 | 12 [10 to 13] | 6.93 [6.14 to 7.83] | 6.02 [5.33 to 6.81]
  B strain, Day 29:Day 1 | 12 [11 to 14] | 6.18 [5.49 to 6.95] | 6.38 [5.66 to 7.18]
  B strain, Day 50:Day 1 | 49 [45 to 54] | 17 [15 to 18] | 16 [15 to 18]
  B strain, Day 209:Day 1 | 13 [12 to 14] | 5.76 [5.26 to 6.3] | 6.15 [5.62 to 6.73]

11. Secondary Outcome: Percentage of Subjects With HI Titers ≥40 Against Homologous Strains, by Vaccine Group
Description: The percentage of subjects demonstrating HI titers ≥40,against homologous strains, at three weeks and six months after vaccination with aTIV or licensed comparator or TIV.
Time Frame: Day 1, Day 29, Day 50, Day 209
Population: Analysis was done on FAS (Persistence)
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (6 to <72 Months) | Comparator TIV (6 to <72 Months) | TIV (6 to <72 Months)
Number analyzed (Participants) | 715 | 822 | 820
Percentage of subjects
  H1N1, Day 1 (N=714,822,820) | 40.6 [37 to 44.3] | 33.1 [29.9 to 36.4] | 36.3 [33 to 39.7]
  H1N1, Day 29 | 89.8 [87.3 to 91.9] | 55 [51.5 to 58.4] | 57.9 [54.5 to 61.3]
  H1N1, Day 50 (N=714,822,820) | 99.3 [98.4 to 99.8] | 91.1 [89 to 93] | 88.2 [85.8 to 90.3]
  H1N1, Day 209 (N=715, 822,819) | 88.8 [86.3 to 91] | 59.5 [56 to 62.9] | 63.2 [59.8 to 66.6]
  H3N2, Day 1 | 52.6 [48.9 to 56.3] | 45.5 [42.1 to 49] | 44.6 [41.2 to 48.1]
  H3N2, Day 29 | 98.9 [97.8 to 99.5] | 95.9 [94.3 to 97.1] | 93.5 [91.6 to 95.1]
  H3N2, Day 50 | 99.7 [99 to 100] | 99.5 [98.8 to 99.9] | 99.4 [98.6 to 99.8]
  H3N2, Day 209 | 99.3 [98.4 to 99.8] | 94.3 [92.5 to 95.8] | 88.4 [86 to 90.5]
  B strain, Day 1 | 22.1 [19.1 to 25.3] | 21.1 [18.3 to 24] | 20.5 [17.8 to 23.4]
  B strain, Day 29 | 69 [65.4 to 72.3] | 48.2 [44.7 to 51.7] | 45.6 [42.2 to 49.1]
  B strain, Day 50 | 98.9 [97.8 to 99.5] | 89.1 [86.7 to 91.1] | 87 [84.5 to 89.2]
  B strain, Day 209 | 93.4 [91.4 to 95.1] | 67.9 [64.6 to 71.1] | 67 [63.6 to 70.2]

12. Secondary Outcome: Percentage of Subjects Achieving Seroconversion or ≥4 Fold Increase in HI Titers, Against Homologous Strains
Description: The percentage of subjects achieving seroconversion ≥4 fold increase in HI titers from baseline, against homologous strains, at three weeks and six months after vaccination with ATIV or licensed comparator or TIV.
Time Frame: Day 29, Day 50, Day 209
Population: Analysis was done on FAS (Persistence)
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (6 to <72 Months) | Comparator TIV (6 to <72 Months) | TIV (6 to <72 Months)
Number analyzed (Participants) | 715 | 822 | 820
Percentage of subjects
  H1N1, Day 29 (N=714,822,820) | 83.6 [80.7 to 86.3] | 48.5 [45.1 to 52.1] | 51.5 [48 to 54.9]
  H1N1, Day 50 (N=713,822,820) | 92.6 [90.4 to 94.4] | 83.9 [81.3 to 86.4] | 79 [76.1 to 81.8]
  H1N1, Day 209 (N=714,822,819) | 71.7 [68.3 to 75] | 39.5 [36.2 to 43] | 41.9 [38.5 to 45.3]
  H3N2, Day 29 | 95.8 [94.1 to 97.2] | 90.3 [88 to 92.2] | 86.7 [84.2 to 89]
  H3N2, Day 50 | 96.5 [94.9 to 97.7] | 92.1 [90 to 93.8] | 90 [87.7 to 92]
  H3N2, Day 209 | 77.6 [74.4 to 80.6] | 62.5 [59.1 to 65.9] | 55.6 [52.1 to 59.1]
  B strain, Day 29 | 68.4 [64.8 to 71.8] | 47 [43.5 to 50.4] | 44 [40.6 to 47.5]
  B strain, Day 50 | 97.6 [96.2 to 98.6] | 86.6 [84.1 to 88.9] | 85 [82.4 to 87.4]
  B strain, Day 209 | 87.3 [84.6 to 89.6] | 59.7 [56.3 to 63.1] | 61.5 [58 to 64.8]

13. Secondary Outcome: Comparison of Antibody Responses of aTIV With TIV and Comparator TIV in Terms of GMTs Against Homologous Strains, Subjects at Risk/Not at Risk, by Age Subgroup
Description: The non-inferiority of Hemagglutination Inhibition (HI) antibody responses of aTIV compared to TIV and comparator TIV assessed in terms of post vaccination GMTs at three weeks after last vaccination against the three homologous vaccine strains, in subjects with a defined set of underlying medical conditions (at risk) and healthy subjects (not at risk), by age sub group.
Time Frame: Day 50
Population: Analysis was done on the PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Compartor TIV (6 to <72 Months): Subjects received a licensed comparator trivalent split influenza vaccine (comparator TIV), subjects aged between 6 to <36 months received two doses (Day 1 & 29) while subjects aged ≥36 months received one dose (at Day 1) of the vaccine
- aTIV (6 to <36 Months): Subjects received two doses (Day 1 & 29) of an investigational MF59-adjuvanted trivalent influenza vaccine (aTIV)
- Compartor TIV (6 to <36 Months): Subjects received two doses (Day 1 & 29) of a licensed comparator trivalent split influenza vaccine (comparator TIV)
- TIV (6 to <36 Months): Subjects received two doses (Day 1 & 29) of an investigational trivalent split influenza vaccine (TIV)
- aTIV (36 to <72 Months): Subjects received one dose (Day 1) of investigational MF59-adjuvanted trivalent influenza vaccine (aTIV)
- Comparator TIV (36 to <72 Months): Subjects received one dose (Day 1) of a licensed comparator trivalent split influenza vaccine (comparator TIV)
- TIV (36 to <72 Months): Subjects received one dose (Day 1) of an investigational trivalent split influenza vaccine (TIV)
Arm/Group | aTIV (6 to <72 Months) | Compartor TIV (6 to <72 Months) | TIV (6 to <72 Months) | aTIV (6 to <36 Months) | Compartor TIV (6 to <36 Months) | TIV (6 to <36 Months) | aTIV (36 to <72 Months) | Comparator TIV (36 to <72 Months) | TIV (36 to <72 Months)
Number analyzed (Participants) | 660 | 722 | 739 | 425 | 612 | 623 | 235 | 110 | 116
Titers
  H1N1nonrisk(N=659,722,739,425,612,623,234,110,116) | 1516 [1358 to 1692] | 566 [509 to 628] | 431 [388 to 478] | 1341 [1165 to 1544] | 478 [425 to 537] | 366 [326 to 411] | 2111 [1840 to 2423] | 1365 [1117 to 1668] | 879 [723 to 1068]
  H3N2nonrisk(N=660,722,739,425,612,623,235,110,116) | 1897 [1772 to 2030] | 1014 [950 to 1082] | 804 [754 to 857] | 1863 [1711 to 2028] | 912 [849 to 979] | 695 [648 to 746] | 2311 [2080 to 2568] | 1526 [1309 to 1780] | 1497 [1289 to 1739]
  B nonrisk(N=660,722,739,425,612,623,235,110,116) | 492 [450 to 539] | 162 [148 to 176] | 157 [144 to 170] | 559 [498 to 627] | 149 [136 to 164] | 141 [128 to 155] | 431 [380 to 488] | 226 [188 to 272] | 254 [212 to 304]
  H1N1 at risk(N=22,35,26,12,23,19,10,12,7) | 1706 [990 to 2939] | 772 [502 to 1185] | 631 [383 to 1041] | 1414 [658 to 3040] | 603 [350 to 1040] | 519 [283 to 950] | 2187 [956 to 5002] | 1241 [583 to 2641] | 1030 [383 to 2767]
  H3N2 at risk(N=22,35,26,12,23,19,10,12,7) | 2306 [1665 to 3194] | 941 [727 to 1220] | 709 [526 to 955] | 2323 [1407 to 3835] | 794 [552 to 1140] | 665 [447 to 988] | 2319 [1622 to 3315] | 1306 [940 to 1815] | 826 [538 to 1267]
  B at risk(N=22,35,26,12,23,19,10,12,7) | 495 [307 to 797] | 143 [98 to 209] | 179 [116 to 278] | 694 [367 to 1316] | 125 [79 to 199] | 132 [79 to 220] | 365 [184 to 724] | 200 [108 to 372] | 312 [131 to 743]
Statistical Analysis 1: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — Noninferiority was concluded if the lower limit of the 2-sided 97.6% confidence interval of the postvaccination (day 50) ratio of GMTs was above 0.667; GMT Ratio (H1N1 strain) = 2.68, 95% CI 2-sided [2.3 to 3.12]
Statistical Analysis 2: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT Ratio (H3N2 strain) = 1.87, 95% CI 2-sided [1.7 to 2.05]
Statistical Analysis 3: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 3.04, 95% CI 2-sided [2.68 to 3.44]
Statistical Analysis 4: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 2.21, 95% CI 2-sided [1.11 to 4.42]
Statistical Analysis 5: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 2.45, 95% CI 2-sided [1.61 to 3.72]
Statistical Analysis 6: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 3.46, 95% CI 2-sided [1.88 to 6.34]
Statistical Analysis 7: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratios (H1N1 strain) = 3.52, 95% CI 2-sided [3.03 to 4.1]
Statistical Analysis 8: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 2.36, 95% CI 2-sided [2.15 to 2.59]
Statistical Analysis 9: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 3.14, 95% CI 2-sided [2.78 to 3.56]
Statistical Analysis 10: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 2.7, 95% CI 2-sided [1.28 to 5.68]
Statistical Analysis 11: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 3.25, 95% CI 2-sided [2.09 to 5.06]
Statistical Analysis 12: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 2.76, 95% CI 2-sided [1.44 to 5.3]
Statistical Analysis 13: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 2.81, 95% CI 2-sided [2.34 to 3.37]
Statistical Analysis 14: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 2.04, 95% CI 2-sided [1.83 to 2.28]
Statistical Analysis 15: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 3.74, 95% CI 2-sided [3.22 to 4.34]
Statistical Analysis 16: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 2.34, 95% CI 2-sided [0.92 to 6]
Statistical Analysis 17: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 2.93, 95% CI 2-sided [1.57 to 5.45]
Statistical Analysis 18: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 5.55, 95% CI 2-sided [2.52 to 12]
Statistical Analysis 19: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 3.66, 95% CI 2-sided [3.05 to 4.39]
Statistical Analysis 20: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 2.68, 95% CI 2-sided [2.4 to 2.99]
Statistical Analysis 21: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 3.97, 95% CI 2-sided [3.42 to 4.61]
Statistical Analysis 22: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 2.72, 95% CI 2-sided [1.02 to 7.31]
Statistical Analysis 23: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 3.5, 95% CI 2-sided [1.85 to 6.62]
Statistical Analysis 24: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 5.26, 95% CI 2-sided [2.32 to 12]
Statistical Analysis 25: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 1.55, 95% CI 2-sided [1.21 to 1.97]
Statistical Analysis 26: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 1.51, 95% CI 2-sided [1.26 to 1.82]
Statistical Analysis 27: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 1.9, 95% CI 2-sided [1.52 to 2.38]
Statistical Analysis 28: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 1.76, 95% CI 2-sided [0.57 to 5.4]
Statistical Analysis 29: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 1.78, 95% CI 2-sided [1.09 to 2.89]
Statistical Analysis 30: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 1.82, 95% CI 2-sided [0.73 to 4.54]
Statistical Analysis 31: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 2.4, 95% CI 2-sided [1.89 to 3.05]
Statistical Analysis 32: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 1.54, 95% CI 2-sided [1.29 to 1.85]
Statistical Analysis 33: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 1.7, 95% CI 2-sided [1.36 to 2.11]
Statistical Analysis 34: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 2.12, 95% CI 2-sided [0.58 to 7.71]
Statistical Analysis 35: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 2.81, 95% CI 2-sided [1.61 to 4.89]
Statistical Analysis 36: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 1.17, 95% CI 2-sided [0.37 to 3.67]

14. Secondary Outcome: Comparison of Antibody Responses of aTIV Versus Comparator TIV and TIV in Terms of Percentage of Subjects Achieving Seroconversion or ≥4-fold Increase in HI Titer Against Homologous Strains in Subjects at Risk/Not at Risk, by Age Subgroup
Description: The non-inferiority of HI antibody responses of aTIV to that of the licensed comparator TIV and to investigational TIV was assessed in terms of percentage of subjects achieving seroconversion or ≥4-fold increase in HI titers at three weeks after last vaccination against the three homologous vaccine strains in subjects with a defined set of underlying medical conditions (at risk) and in healthy subjects (not at risk) , by age sub group.
Time Frame: Day 50
Population: Analysis was done on the Per Protocol Set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | aTIV (6 to <72 Months) | Compartor TIV (6 to <72 Months) | TIV (6 to <72 Months) | aTIV (6 to <36 Months) | Compartor TIV (6 to <36 Months) | TIV (6 to <36 Months) | aTIV (36 to <72 Months) | Comparator TIV (36 to <72 Months) | TIV (36 to <72 Months)
Number analyzed (Participants) | 660 | 722 | 739 | 425 | 612 | 623 | 235 | 110 | 116
Percentages of subjects
  H1N1 norisk(N=658,722,739,425,612,623,233,110,116) | 93 [91 to 95] | 85 [82 to 87] | 79 [76 to 82] | 95 [92 to 97] | 84 [81 to 87] | 78 [75 to 82] | 91 [86 to 94] | 88 [81 to 94] | 83 [75 to 89]
  H3N2 norisk(N=660,722,739,425,612,623,235,110,116) | 97 [95 to 98] | 93 [91 to 94] | 90 [87 to 92] | 98 [96 to 99] | 93 [91 to 95] | 90 [88 to 93] | 94 [91 to 97] | 90 [83 to 95] | 86 [79 to 92]
  B norisk(N=660,722,739,425,612,623,235,110,116) | 98 [96 to 99] | 86 [83 to 88] | 84 [82 to 87] | 98 [96 to 99] | 85 [82 to 88] | 83 [79 to 86] | 98 [95 to 99] | 90 [83 to 95] | 94 [88 to 98]
  H1N1 at risk (N=22,35,26,12,23,19,10,12,7) | 82 [60 to 95] | 83 [66 to 93] | 85 [65 to 96] | 92 [62 to 100] | 87 [66 to 97] | 89 [67 to 99] | 70 [35 to 93] | 75 [43 to 95] | 71 [29 to 96]
  H3N2 at risk(N=22,35,26,12,23,19,10,12,7) | 86 [65 to 97] | 86 [70 to 95] | 81 [61 to 93] | 83 [52 to 98] | 78 [56 to 93] | 74 [49 to 91] | 90 [55 to 100] | 100 [74 to 100] | 100 [59 to 100]
  B at risk(N=22,35,26,12,23,19,10,12,7) | 100 [85 to 100] | 86 [70 to 98] | 88 [70 to 98] | 100 [74 to 100] | 91 [72 to 99] | 84 [60 to 97] | 100 [69 to 100] | 75 [43 to 95] | 100 [59 to 100]
Statistical Analysis 1: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the lower bound of confidence interval for day 50 vaccine group difference was > -10%; Group difference (H1N1 strain) = 9, 95% CI 2-sided [5.4 to 12]
Statistical Analysis 2: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 4, 95% CI 2-sided [1.8 to 6.6]
Statistical Analysis 3: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 12, 95% CI 2-sided [9.2 to 14.8]
Statistical Analysis 4: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = -1, 95% CI 2-sided [-24 to 18.7]
Statistical Analysis 5: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 1, 95% CI 2-sided [-21.2 to 18.9]
Statistical Analysis 6: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 14, 95% CI 2-sided [-1.6 to 29.5]
Statistical Analysis 7: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = 14, 95% CI 2-sided [10.7 to 17.7]
Statistical Analysis 8: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 7, 95% CI 2-sided [4.6 to 9.8]
Statistical Analysis 9: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 13, 95% CI 2-sided [10.7 to 16.4]
Statistical Analysis 10: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = -3, 95% CI 2-sided [-26.1 to 19.2]
Statistical Analysis 11: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 6, 95% CI 2-sided [-17.5 to 27.3]
Statistical Analysis 12: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 12, 95% CI 2-sided [-4.4 to 29.2]
Statistical Analysis 13: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = 11, 95% CI 2-sided [7.2 to 14.5]
Statistical Analysis 14: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 5, 95% CI 2-sided [2.6 to 7.5]
Statistical Analysis 15: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 13, 95% CI 2-sided [9.5 to 15.8]
Statistical Analysis 16: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = 5, 95% CI 2-sided [-24.7 to 26.3]
Statistical Analysis 17: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 5, 95% CI 2-sided [-26.9 to 30.3]
Statistical Analysis 18: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 9, 95% CI 2-sided [-16.9 to 27.1]
Statistical Analysis 19: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = 16, 95% CI 2-sided [12.4 to 20.2]
Statistical Analysis 20: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 8, 95% CI 2-sided [5.1 to 10.5]
Statistical Analysis 21: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 15, 95% CI 2-sided [12 to 18.6]
Statistical Analysis 22: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = 2, 95% CI 2-sided [-27.1 to 25.5]
Statistical Analysis 23: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 10, 95% CI 2-sided [-23.5 to 37.2]
Statistical Analysis 24: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 16, 95% CI 2-sided [-10.7 to 38]
Statistical Analysis 25: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = 2, 95% CI 2-sided [-4.2 to 10.4]
Statistical Analysis 26: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 subjects) = 4, 95% CI 2-sided [-1.2 to 11.9]
Statistical Analysis 27: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 8, 95% CI 2-sided [2.9 to 15.1]
Statistical Analysis 28: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = -5, 95% CI 2-sided [-42.4 to 32]
Statistical Analysis 29: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = -10, 95% CI 2-sided [-41.2 to 16.6]
Statistical Analysis 30: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 25, 95% CI 2-sided [-7.1 to 53.9]
Statistical Analysis 31: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = 8, 95% CI 2-sided [1 to 16.4]
Statistical Analysis 32: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 8, 95% CI 2-sided [2 to 16.1]
Statistical Analysis 33: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 4, 95% CI 2-sided [0 to 10]
Statistical Analysis 34: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = -1, 95% CI 2-sided [-42.1 to 43]
Statistical Analysis 35: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = -10, 95% CI 2-sided [-41.5 to 28.7]
Statistical Analysis 36: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 0, 95% CI 2-sided [-29 to 36.8]

15. Secondary Outcome: Comparison of Antibody Responses of TIV Versus Comparator TIV in Terms of Percentage of Subjects Achieving Seroconversion or ≥4-fold Increase in HI Titer Against Homologous Strains in Subjects at Risk/Not at Risk, by Age Sub Group-FAS
Description: The superiority of HI antibody responses of aTIV compared to TIV and comparator TIV assessed in terms of of percentage of subjects achieving seroconversion or ≥4-fold increase in HI Titer at three weeks after last vaccination against the three homologous vaccine strains in subjects with a defined set of underlying medical conditions (at risk) and healthy subjects (not at risk), by age sub group.
Time Frame: Day 50
Population: Analysis was done on the Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | aTIV (6 to <72 Months) | Compartor TIV (6 to <72 Months) | TIV (6 to <72 Months) | aTIV (6 to <36 Months) | Compartor TIV (6 to <36 Months) | TIV (6 to <36 Months) | aTIV (36 to <72 Months) | Comparator TIV (36 to <72 Months) | TIV (36 to <72 Months)
Number analyzed (Participants) | 719 | 799 | 814 | 459 | 673 | 688 | 260 | 126 | 126
Percentages of subjects
  H1N1 norisk(N=717,799,814,459,673,688,258,126,126) | 93 [91 to 95] | 84 [81 to 86] | 79 [76 to 81] | 95 [92 to 96] | 83 [80 to 86] | 78 [75 to 81] | 91 [87 to 94] | 89 [82 to 94] | 81 [73 to 87]
  H3N2 norisk(N=719,799,814,459,673,688,260,126,126) | 97 [95 to 98] | 93 [91 to 94] | 90 [88 to 92] | 98 [96 to 99] | 93 [91 to 95] | 91 [88 to 93] | 95 [91 to 97] | 91 [85 to 96] | 87 [79 to 92]
  B norisk(N=719,799,814,459,673,688,260,126,126) | 97 [96 to 99] | 86 [84 to 89] | 84 [82 to 87] | 98 [96 to 99] | 85 [83 to 88] | 83 [80 to 85] | 97 [95 to 99] | 91 [85 to 96] | 94 [88 to 97]
  H1N1 at risk(N=28,40,35,17,26,26,11,14,9) | 79 [59 to 92] | 83 [67 to 93] | 83 [66 to 93] | 82 [57 to 96] | 85 [65 to 96] | 85 [65 to 96] | 73 [39 to 94] | 79 [49 to 95] | 78 [40 to 97]
  H3N2 at risk(N=28,40,35,17,26,26,11,14,9) | 89 [72 to 98] | 85 [70 to 94] | 83 [66 to 93] | 88 [64 to 99] | 77 [56 to 91] | 77 [56 to 91] | 91 [59 to 100] | 100 [77 to 100] | 100 [66 to 100]
  B at risk(N=28,40,35,17,26,26,11,14,9) | 96 [82 to 100] | 88 [73 to 96] | 89 [73 to 97] | 94 [71 to 100] | 92 [75 to 99] | 85 [65 to 96] | 100 [72 to 100] | 79 [49 to 95] | 100 [66 to 100]
Statistical Analysis 1: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = 10, 95% CI 2-sided [6.4 to 12.8]
Statistical Analysis 2: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 4, 95% CI 2-sided [1.8 to 6.4]
Statistical Analysis 3: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 11, 95% CI 2-sided [8.6 to 13.9]
Statistical Analysis 4: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = -4, 95% CI 2-sided [-24.7 to 14.9]
Statistical Analysis 5: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 4, 95% CI 2-sided [-14.4 to 20.7]
Statistical Analysis 6: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 9, 95% CI 2-sided [-6.8 to 23.4]
Statistical Analysis 7: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = 15, 95% CI 2-sided [11.3 to 18.1]
Statistical Analysis 8: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 7, 95% CI 2-sided [4.2 to 9.1]
Statistical Analysis 9: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 13, 95% CI 2-sided [10.5 to 16.1]
Statistical Analysis 10: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = -4, 95% CI 2-sided [-25.3 to 15.4]
Statistical Analysis 11: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 6, 95% CI 2-sided [-12.7 to 24.2]
Statistical Analysis 12: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group differences (B strain) = 8, 95% CI 2-sided [-7.8 to 23.2]
Statistical Analysis 13: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = 12, 95% CI 2-sided [8.2 to 15.3]
Statistical Analysis 14: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 5, 95% CI 2-sided [2.5 to 7.4]
Statistical Analysis 15: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 12, 95% CI 2-sided [9.2 to 15.3]
Statistical Analysis 16: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = -2, 95% CI 2-sided [-28.5 to 20.2]
Statistical Analysis 17: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 11, 95% CI 2-sided [-14.9 to 33.5]
Statistical Analysis 18: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 2, 95% CI 2-sided [-20.7 to 19.7]
Statistical Analysis 19: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = 16, 95% CI 2-sided [12.6 to 20.1]
Statistical Analysis 20: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 7, 95% CI 2-sided [4.6 to 9.8]
Statistical Analysis 21: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 15, 95% CI 2-sided [11.9 to 18.3]
Statistical Analysis 22: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = -2, 95% CI 2-sided [-28.5 to 20.2]
Statistical Analysis 23: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 11, 95% CI 2-sided [-14.9 to 33.5]
Statistical Analysis 24: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 10, 95% CI 2-sided [-14 to 29.3]
Statistical Analysis 25: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = 2, 95% CI 2-sided [-3.8 to 9.5]
Statistical Analysis 26: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 3, 95% CI 2-sided [-1.8 to 10]
Statistical Analysis 27: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 6, 95% CI 2-sided [1.5 to 12.5]
Statistical Analysis 28: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = -6, 95% CI 2-sided [-40.7 to 27.9]
Statistical Analysis 29: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = -9, 95% CI 2-sided [-38.4 to 14.3]
Statistical Analysis 30: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 21, 95% CI 2-sided [-7.9 to 48.1]
Statistical Analysis 31: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = 10, 95% CI 2-sided [3 to 18.5]
Statistical Analysis 32: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = 8, 95% CI 2-sided [2.2 to 15.6]
Statistical Analysis 33: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 4, 95% CI 2-sided [0 to 9.6]
Statistical Analysis 34: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H1N1 strain) = -5, 95% CI 2-sided [-41.7 to 35]
Statistical Analysis 35: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (H3N2 strain) = -9, 95% CI 2-sided [-38.6 to 23.4]
Statistical Analysis 36: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; Group difference (B strain) = 0, 95% CI 2-sided [-26.9 to 31]

16. Secondary Outcome: Comparison of Antibody Responses of aTIV With TIV and Comparator TIV in Terms of GMTs Against Homologous Strains, at Risk/Not at Risk, by Age Sub Group-FAS
Description: The superiority of HI antibody responses of aTIV compared to TIV and comparator TIV assessed in terms of post vaccination GMTs at three weeks after last vaccination against the three homologous vaccine strains, in subjects with a defined set of underlying medical conditions (at risk) and in healthy subjects (not at risk), by age sub group.
Time Frame: Day 50
Population: Analysis was done on Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | aTIV (6 to <72 Months) | Compartor TIV (6 to <72 Months) | TIV (6 to <72 Months) | aTIV (6 to <36 Months) | Compartor TIV (6 to <36 Months) | TIV (6 to <36 Months) | aTIV (36 to <72 Months) | Comparator TIV (36 to <72 Months) | TIV (36 to <72 Months)
Number analyzed (Participants) | 719 | 799 | 814 | 459 | 673 | 688 | 260 | 126 | 126
Titers
  H1N1 norisk(N=718,799,814,459,673,688,259,126,126) | 1509 [1357 to 1677] | 569 [515 to 629] | 422 [382 to 466] | 1336 [1166 to 1530] | 474 [424 to 530] | 365 [326 to 407] | 2077 [1815 to 2376] | 1413 [1165 to 1713] | 813 [670 to 986]
  H3N2 norisk(N=719,799,814,459,673,688,260,126,126) | 1894 [1775 to 2022] | 1015 [954 to 1080] | 794 [747 to 844] | 1851 [1705 to 2010] | 905 [845 to 968] | 686 [641 to 733] | 2343 [2120 to 2589] | 1582 [1370 to 1826] | 1475 [1278 to 1703]
  B norisk(N=719,799,814,459,673,688,260,126,126) | 484 [444 to 527] | 164 [151 to 178] | 155 [143 to 168] | 545 [487 to 608] | 150 [137 to 164] | 139 [127 to 152] | 432 [383 to 487] | 243 [205 to 289] | 253 [212 to 300]
  H1N1 at risk(N=28,40,35,17,26,26,11,14,9) | 1541 [948 to 2504] | 830 [553 to 1244] | 586 [380 to 905] | 1277 [674 to 2418] | 617 [370 to 1028] | 483 [289 to 808] | 1982 [929 to 4228] | 1478 [756 to 2891] | 1028 [445 to 2372]
  H3N2 at risk(N=28,40,35,17,26,26,11,14,9) | 2361 [1743 to 3197] | 960 [744 to 1237] | 763 [582 to 1001] | 2517 [1633 to 3881] | 820 [578 to 1164] | 705 [496 to 1000] | 2197 [1514 to 3187] | 1286 [925 to 1788] | 929 [616 to 1399]
  B at risk(N=28,40,35,17,26,26,11,14,9) | 399 [254 to 628] | 152 [104 to 222] | 183 [122 to 274] | 508 [274 to 939] | 140 [85 to 231] | 147 [89 to 242] | 319 [170 to 596] | 197 [114 to 341] | 241 [118 to 493]
Statistical Analysis 1: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT Ratio (H1N1 strain) = 2.29, 95% CI 2-sided [1.91 to 2.76]
Statistical Analysis 2: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT Ratio (H3N2 strain) = 1.6, 95% CI 2-sided [1.35 to 1.89]
Statistical Analysis 3: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 2.92, 95% CI 2-sided [2.57 to 3.31]
Statistical Analysis 4: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 1.53, 95% CI 2-sided [0.6 to 3.93]
Statistical Analysis 5: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 2.02, 95% CI 2-sided [0.89 to 4.61]
Statistical Analysis 6: Comparison: aTIV (6 to <72 Months) vs Compartor TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 2.5, 95% CI 2-sided [1.34 to 4.67]
Statistical Analysis 7: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 3.33, 95% CI 2-sided [2.77 to 4.01]
Statistical Analysis 8: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 2.07, 95% CI 2-sided [1.75 to 2.45]
Statistical Analysis 9: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 3.08, 95% CI 2-sided [2.72 to 3.49]
Statistical Analysis 10: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 1.71, 95% CI 2-sided [0.65 to 4.5]
Statistical Analysis 11: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 3.22, 95% CI 2-sided [1.38 to 7.51]
Statistical Analysis 12: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 2.1, 95% CI 2-sided [1.1 to 3.98]
Statistical Analysis 13: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; GMT ratio (H1N1 strain) = 2.59, 95% CI 2-sided [2.1 to 3.21]
Statistical Analysis 14: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; GMT ratio (H3N2 strain) = 2.08, 95% CI 2-sided [1.71 to 2.52]
Statistical Analysis 15: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; GMT ratio (B strain) = 3.73, 95% CI 2-sided [3.22 to 4.33]
Statistical Analysis 16: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; GMT ratio (H1N1 strain) = 1.4, 95% CI 2-sided [0.45 to 4.4]
Statistical Analysis 17: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; GMT ratio (H3N2 strain) = 2.86, 95% CI 2-sided [0.94 to 8.66]
Statistical Analysis 18: Comparison: aTIV (6 to <36 Months) vs Compartor TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; GMT ratio (B strain) = 1.4, 95% CI 2-sided [0.45 to 4.4]
Statistical Analysis 19: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; GMT ratio (H1N1 strain) = 3.67, 95% CI 2-sided [2.97 to 4.54]
Statistical Analysis 20: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; GMT ratio (H3N2 strain) = 2.78, 95% CI 2-sided [2.29 to 3.37]
Statistical Analysis 21: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; GMT ratio (B strain) = 4.01, 95% CI 2-sided [3.46 to 4.65]
Statistical Analysis 22: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 14, analysis 1]; GMT ratio (H1N1 strain) = 1.4, 95% CI 2-sided [0.45 to 4.4]
Statistical Analysis 23: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 4.32, 95% CI 2-sided [1.43 to 13]
Statistical Analysis 24: Comparison: aTIV (6 to <36 Months) vs TIV (6 to <36 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 3.69, 95% CI 2-sided [1.67 to 8.15]
Statistical Analysis 25: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 1.35, 95% CI 2-sided [0.89 to 2.04]
Statistical Analysis 26: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 1.59, 95% CI 2-sided [1.14 to 2.22]
Statistical Analysis 27: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 1.68, 95% CI 2-sided [1.3 to 2.15]
Statistical Analysis 28: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 1.73, 95% CI 2-sided [0.29 to 10]
Statistical Analysis 29: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 1.16, 95% CI 2-sided [0.33 to 4.01]
Statistical Analysis 30: Comparison: aTIV (36 to <72 Months) vs Comparator TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 1.45, 95% CI 2-sided [0.53 to 3.94]
Statistical Analysis 31: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 2.24, 95% CI 2-sided [1.48 to 3.39]
Statistical Analysis 32: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 1.76, 95% CI 2-sided [1.26 to 2.46]
Statistical Analysis 33: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); No risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 1.59, 95% CI 2-sided [1.24 to 2.04]
Statistical Analysis 34: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H1N1 strain) = 2.48, 95% CI 2-sided [0.34 to 18]
Statistical Analysis 35: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (H3N2 strain) = 1.98, 95% CI 2-sided [0.49 to 7.92]
Statistical Analysis 36: Comparison: aTIV (36 to <72 Months) vs TIV (36 to <72 Months); At risk subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; GMT ratio (B strain) = 0.71, 95% CI 2-sided [0.23 to 2.16]

17. Secondary Outcome: The HI GMTs Against Heterologous Strains, by Vaccine Group (6 to <72 Months Age Group)
Description: The HI antibody titers against the heterologous strains following vaccination with either aTIV, licensed comparator or TIV, at three weeks and at six months after vaccination are reported as GMTs.
Time Frame: Day 1, Day 50, Day 209
Population: Analysis was done on the FAS Persistence
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | aTIV (6 to <72 Months) | Comparator TIV (6 to <72 Months) | TIV (6 to <72 Months)
Number analyzed (Participants) | 380 | 445 | 431
Titers
  H1N1/Jersey - Day 1 (N=380,445,430) | 10 [9.37 to 11] | 9.75 [8.85 to 11] | 10 [9.07 to 11]
  H1N1/Jersey - Day 50 | 51 [45 to 58] | 29 [26 to 33] | 31 [27 to 36]
  H1N1/Jersey - Day 209 | 21 [19 to 23] | 17 [16 to 19] | 18 [16 to 20]
  H3N2/Uruguay - Day 1 (N=380,445,430) | 17 [15 to 20] | 18 [16 to 20] | 17 [15 to 19]
  H3N2/Uruguay - Day 50 | 184 [165 to 206] | 88 [79 to 98] | 71 [63 to 79]
  H3N2/Uruguay- Day 209 | 42 [37 to 47] | 31 [28 to 34] | 27 [24 to 30]
  B strain - Day 1 | 5.98 [5.72 to 6.25] | 5.8 [5.55 to 6.05] | 5.85 [5.6 to 6.11]
  B strain - Day 50 | 99 [89 to 111] | 34 [31 to 38] | 35 [31 to 39]
  B strain Day 209 | 20 [18 to 22] | 11 [9.86 to 12] | 11 [9.94 to 12]

18. Secondary Outcome: Percentage of Subjects Achieving Seroconversion or ≥4 Fold Increase in HI Titers, Against Heterologous Strains
Description: The percentage of subjects achieving seroconversion or ≥4 fold increase in HI titers from baseline, against heterologous strains, at three weeks and six months after last vaccination with aTIV or licensed comparator or TIV.
Time Frame: Day 50, Day 209
Population: Subjects aged 6 through <72 months of age - Full Analyses Set (FAS) Persistence
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (6 to <72 Months) | Comparator TIV (6 to <72 Months) | TIV (6 to <72 Months)
Number analyzed (Participants) | 380 | 445 | 431
Percentage of subjects
  H1N1/Jersey, Day 50 (N=380,445,430) | 53.16 [48.00 to 58.26] | 36.85 [32.36 to 41.52] | 36.05 [31.50 to 40.78]
  H1N1/Jersey, Day 209 (N=380,445,430) | 33.95 [29.20 to 38.95] | 19.33 [15.76 to 23.31] | 20.70 [16.96 to 24.84]
  H3N2/Uruguay, Day 50 (N=380,445,430) | 91.84 [88.62 to 94.39] | 60.9 [56.19 to 65.46] | 53.26 [48.42 to 58.05]
  H3N2/Uruguay, Day 209 (N=380,445,430) | 40.26 [35.29 to 45.39] | 23.82 [19.94 to 28.06] | 19.07 [15.46 to 23.11]
  B strain, Day 50 | 92.63 [89.53 to 95.05] | 53.71 [48.95 to 58.41] | 52.90 [48.07 to 57.69]
  B strain, Day 209 | 30.0 [25.43 to 34.88] | 13.93 [10.85 to 17.50] | 17.63 [14.15 to 21.57]

19. Secondary Outcome: Comparison of Antibody Responses of aTIV With TIV and Comparator TIV in Terms of GMTs Against Homologous Strains, After One Vaccination
Description: To demonstrate the GMTs at three weeks after one dose of aTIV are statistically significantly higher to the corresponding response's of comparator TIV and TIV.
Time Frame: Day 1, Day 29
Population: Analysis was done on the FAS (Persistence).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | aTIV (6 to <72 Months) | Comparator TIV (6 to <72 Months) | TIV (6 to <72 Months)
Number analyzed (Participants) | 715 | 822 | 820
Titers
  H1N1- Day 1 (N=714,822,820) | 28 [24 to 32] | 24 [20 to 27] | 27 [23 to 31]
  H1N1- Day 29 | 647 [562 to 745] | 159 [139 to 182] | 170 [148 to 194]
  H3N2 - Day 1 | 42 [36 to 48] | 43 [37 to 49] | 43 [38 to 50]
  H3N2 - Day 29 | 1087 [1004 to 1176] | 558 [517 to 602] | 453 [420 to 490]
  B strain Day 1 | 10 [9.29 to 11] | 10 [9.57 to 11] | 10 [9.34 to 11]
  B strain Day 29 | 119 [106 to 134] | 58 [52 to 65] | 61 [54 to 68]
Statistical Analysis 1: Comparison: aTIV (6 to <72 Months) vs Comparator TIV (6 to <72 Months); GMTs were considered to be statistically significantly higher if the lower bound of the 95% confidence interval around the vaccine group ratio was >1.0; Test type: Superiority or Other; GMT ratio (H1N1 strain) = 4.07, 95% CI 2-sided [3.34 to 4.95]
Statistical Analysis 2: Comparison: aTIV (6 to <72 Months) vs Comparator TIV (6 to <72 Months); statistically significantly greater response was concluded if the lower bound of the 95% confidence interval around the vaccine group ratio is >1.0; Test type: Superiority or Other; GMT ratio (H3N2 strain) = 1.95, 95% CI 2-sided [1.74 to 2.18]
Statistical Analysis 3: Comparison: aTIV (6 to <72 Months) vs Comparator TIV (6 to <72 Months); statistically significantly greater response was concluded if the lower bound of the 95% CI around the vaccine group ratio was >1.0; Test type: Superiority or Other; GMT ratio (B strain) = 2.03, 95% CI 2-sided [1.73 to 2.39]
Statistical Analysis 4: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; GMT ratio (H1N1 strain) = 3.82, 95% CI [3.14 to 4.64]
Statistical Analysis 5: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; GMT ratio (H3N2 strain) = 2.4, 95% CI 2-sided [2.15 to 2.68]
Statistical Analysis 6: Comparison: aTIV (6 to <72 Months) vs TIV (6 to <72 Months); [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; GMT ratio (B strain) = 1.95, 95% CI 2-sided [1.65 to 2.29]

20. Secondary Outcome: Number of Subjects Reporting Solicited Adverse Events After Vaccination
Description: The number of subjects reporting any solicited local and systemic adverse events (AEs), following vaccination with aTIV or licensed comparator or TIV.
Time Frame: Day 1 through Day 7 after any vaccination
Population: Analysis was done on solicited safety set i.e all subjects who had received at least one study vaccine and had provided data on post vaccination solicited AEs
Measure: Number; unit: Participants
Arm/Group | aTIV (6 to <72 Months) | TIV (6 to <72 Months) | Comparator TIV (6 to <72 Months)
Number analyzed (Participants) | 3082 | 1453 | 1451
Participants
  Any local | 1082 | 292 | 311
  Injection site ecchymosis(N=3075,1450,1446) | 191 | 72 | 86
  Injection site erythema (N=3075,1450,1446) | 312 | 109 | 101
  Injection site induration (N=3075,1450,1446) | 258 | 62 | 67
  Injection site tenderness (N=1495,1025,1012) | 152 | 70 | 78
  Injection site swelling (N=3075,1450,1446) | 217 | 1450 | 1446
  Injection site pain (N=1580,422,429) | 1580 | 422 | 429
  Any systemic | 1487 | 604 | 569
  chills (N=1578,423,428) | 154 | 23 | 18
  Myalgia (N=1578,423,429) | 216 | 43 | 25
  Arthralgia (N=1578,423,429) | 125 | 20 | 16
  Headache (N=1578,423,429) | 282 | 46 | 38
  Fatigue (N=1578,423,430) | 204 | 43 | 31
  Eating Habit (N=3076,1450,1446) | 437 | 196 | 205
  Diarrhea (N=3075,1450,1447) | 423 | 231 | 220
  Irritability (N=1496,1024,1013) | 290 | 164 | 190
  Crying (N=1463,1001,990) | 186 | 105 | 122
  Sleepiness (N=1495,1024,1012) | 229 | 150 | 153
  Vomiting (N=3075,1451,1446) | 249 | 100 | 104
  Fever (≥38°C) (N=3074,1450,1446) | 748 | 236 | 224
  Any other | 1047 | 310 | 317
  Axillary Temperature (≥40°C) (N=3074,1450,1446) | 8 | 4 | 3
  Analgesic Antipyretic Med. used(N=3076,1448,1444) | 984 | 285 | 282

21. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Vaccination
Description: The number of subjects reporting any unsolicited adverse events (AEs) between Day 1 to Day 50, serious adverse events (SAEs), AE leading to withdrawal (WD), new onset of chronic disease(NOCD), adverse events of special interest following vaccination with aTIV or licensed comparator or TIV throughout the study (Day 1 to Day 394).
Time Frame: Day 1 to Day 394
Population: Analysis was done on the safety population i.e all subjects who had received at least one study vaccine and had postvaccination safety data
Measure: Number; unit: Participants
Arm/Group | aTIV (6 to <72 Months) | Comparator TIV (6 to <72 Months) | TIV (6 to <72 Months)
Number analyzed (Participants) | 3123 | 1474 | 1477
Participants
  Any AEs (Day 1 to Day 50) | 1541 | 859 | 808
  Possibly/probably related AEs(Day 1 to Day 50) | 158 | 101 | 84
  Any SAEs | 115 | 64 | 69
  Possibly/probably related SAE | 1 | 0 | 0
  AE leading to WD | 1 | 5 | 4
  NOCD | 48 | 31 | 24
  AESI | 1 | 0 | 0
  Deaths | 1 | 3 | 4

ADVERSE EVENTS:
Time Frame: Solicited AEs collected from Day 1-7 after each vaccination, Unsolicited AEs, Adverse Events of Special Interest, New onset chronic disease, AEs leading to withdrawal and serious adverse events reported for through out the study (Day 1-Day 394)
Description: Analysis was done on Full Safety Set - Subjects who received at least one study vaccination and provided post baseline safety data.
Arm/Group | ATIV (6 to <72 Months) | TIV (6 to <72 Months) | Comparator TIV (6 to <72 Months)
Serious Adverse Events (participants affected / at risk) | 115/3123 | 69/1477 | 64/1474
Other Adverse Events (participants affected / at risk) | 2106/3123 | 905/1477 | 917/1474
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATIV (6 to <72 Months) (N=3123) | TIV (6 to <72 Months) (N=1477) | Comparator TIV (6 to <72 Months) (N=1474)
Coeliac Disease (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Upper Gastrointestinal Disorder Hamorrage (Gastrointestinal disorders) | 0 | 0 | 1
Drowning (General disorders) | 0 | 0 | 1
Type III Immune Complex Mediated Reaction (Immune system disorders) | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 2 | 0
Abscess Limb (Infections and infestations) | 0 | 1 | 0
Abscess Neck (Infections and infestations) | 0 | 1 | 0
Amoebiasis (Infections and infestations) | 1 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 1
Arthritis Bacterial (Infections and infestations) | 0 | 0 | 1
Bacterial Infection (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1
Bronchopneumonia (Infections and infestations) | 4 | 3 | 6
Cellulitis (Infections and infestations) | 0 | 1 | 1
Dengue Fever (Infections and infestations) | 5 | 8 | 3
Diarrhoea Infectious (Infections and infestations) | 0 | 0 | 1
Dysentery (Infections and infestations) | 0 | 1 | 1
Encephalitis Viral (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 18 | 10 | 12
Hepatitis A (Infections and infestations) | 0 | 0 | 1
Lower Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0
Measles (Infections and infestations) | 1 | 0 | 0
Meningitis Pneumococcal (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0
Otitis Media (Infections and infestations) | 1 | 1 | 0
Otitis Media Bacterial (Infections and infestations) | 1 | 0 | 0
Otitis Media Chronic (Infections and infestations) | 1 | 0 | 0
Parasitic Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 26 | 12 | 13
Pneumonia Bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia Viral (Infections and infestations) | 1 | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 1 | 0 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 | 0 | 1
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2
Septic Shock (Infections and infestations) | 1 | 0 | 0
Shigella Infection (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 2 | 1 | 0
Tooth Abscess (Infections and infestations) | 1 | 0 | 0
Thypoid Fever (Infections and infestations) | 1 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 2 | 3
Varicella (Infections and infestations) | 1 | 0 | 0
Viral Infection (Infections and infestations) | 2 | 0 | 2
Viral Rash (Infections and infestations) | 0 | 1 | 0
Accidental Exposure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Animal Bite (Injury, poisoning and procedural complications) | 22 | 15 | 14
Animal Scratch (Injury, poisoning and procedural complications) | 3 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Eye Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Forearm Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skull Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Tetany (Metabolism and nutrition disorders) | 0 | 0 | 1
Acute Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 2 | 0
Febrile Convulsion (Nervous system disorders) | 13 | 4 | 3
Adenoidal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Tonsillary Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Finger Amputation (Surgical and medical procedures) | 1 | 0 | 0
Roseola (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATIV (6 to <72 Months) (N=3123) | TIV (6 to <72 Months) (N=1477) | Comparator TIV (6 to <72 Months) (N=1474)
Diarrhea (Gastrointestinal disorders) | 445 | 247 | 231
Vomiting (Gastrointestinal disorders) | 257 | 107 | 109
Crying (General disorders) | 186 | 105 | 124
Fatigue (General disorders) | 204 | 43 | 31
Injection site erythema (General disorders) | 312 | 109 | 102
Injection site hemorrhage (General disorders) | 191 | 72 | 86
Injection site induration (General disorders) | 258 | 62 | 67
Injection site pain (General disorders) | 851 | 177 | 189
Injection site swelling (General disorders) | 217 | 34 | 43
Irritability postvaccinal (General disorders) | 290 | 165 | 191
Pyrexia (General disorders) | 795 | 279 | 260
Gastroenteritis (Infections and infestations) | 112 | 70 | 84
Nasopharyngitis (Infections and infestations) | 291 | 151 | 175
Upper respiratory tract infection (Infections and infestations) | 452 | 237 | 246
Decreased appetite (Metabolism and nutrition disorders) | 437 | 197 | 206
Myalgia (Musculoskeletal and connective tissue disorders) | 216 | 43 | 25
Headache (Nervous system disorders) | 286 | 48 | 40
Hypersomnia (Nervous system disorders) | 229 | 150 | 153

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days